# Evaluation of the Performance of CONTOUR NEXT® and CONTOUR PLUS ELITE® Blood Glucose Monitoring Systems in Neonates using Capillary Blood Samples

# **Protocol/Clinical Investigation Plan:**

GCA-PRO-2021-003-01

Amendment 1: 14 October 2022

Sponsor: Ascensia Diabetes Care

100 Summit Lake Drive Valhalla, NY 10595



Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1

Version: 140ct2022

Ascensia Diabetes Care

#### **Investigator Statement**

I have read this protocol and agree to conduct the clinical performance study according to the protocol. I understand and agree that before seeking approval from an Institutional Review Board (IRB), the Ascensia Diabetes Care study manager must approve any changes to the protocol. I also agree to protect the rights, safety, dignity, and well-being of the subjects.

Principal Investigator (PI): Dennis Dietzen, PhD

Site: St. Louis Children's Hospital, Washington University

Address: 1 Children's Place

St. Louis, MO 63110

PI Sgnature Printed Name Date

This protocol and the data obtained from the study are confidential and may not be disclosed without the prior written consent of Ascensia Diabetes Care (ADC).

# **Table of Contents**

| Abbr | eviations 5 |
|---|---|
| 1.0 | Identification of the Protocol/ Clinical Investigation Plan (CIP) 6 |
| 2.0 | Contact Information |
| 3.0 | Synopsis of the Clinical Study 8 |
| 4.0 | Identification and description of the investigational device9 |
| 5.0 | Justification for the Design of the Clinical Study10 |
| 6.0 | Risks and benefits of the investigational device and clinical investigation11 |
| 7.0 | Objectives and Hypotheses12 |
| 8.0 | Clinical Study Design |
| 9.0 | Investigational device(s) and comparator(s)13 |
| 10.0 | Subjects14 |
| 11.0 | Procedures15 |
| 12.0 | Monitoring Plan20 |
| 13.0 | Statistical Plan20 |
| 14.0 | Data Management24 |
| 15.0 | Amendments to the Protocol24 |
| 16.0 | Deviations from the clinical protocol26 |

| 17.0 | Device Accountability26 |
|---|---|
| 18.0 | Regulatory27 |
| 19.0 | Statements of compliance28 |
| 20.0 | Informed Consent Process28 |
| 21.0 | Adverse events and adverse device effects29 |
| 22.0 | Handling and Reporting of Device Deficiencies31 |
| 23.0 | Vulnerable population32 |
| 24.0 | Suspension/Premature termination and Subject Withdrawal Criteria32 |
| 25.0 | Results Handling32 |
| 26.0 | Publication policy32 |
| 27.0 | Administration33 |
| 28.0 | Bibliography33 |
| Appen | dix A - Instructions for Cleaning and Disinfecting Meters34 |
| Appen | dix B - Instructions for Processing of Blood for the glucose analyzer35 |
| Appen | dix C - Instructions for Tracking Accuracy and Precision of the Laboratory Glucose Analyzer 36 |
| Appen | dix D - Instructions for Hematocrit Sample Preparation and Testing38 |
| Attach | ment 1 - CONTOUR NEXT User Guide39 |
| Attach | ment 2 - CONTOUR PLUS ELITE User Guide41 |


#### **Abbreviations**

**ADC** Ascensia Diabetes Care

**AE** Adverse Event

**ADE** Adverse Device Effect

**BG** Blood Glucose

**BGMS** Blood Glucose Monitoring System

CIP Clinical Investigation Plan (Protocol)

**CRF** Case Report Form

**EDC** Electronic Data Capture

**GCP** Good Clinical Practice

**HCP** Health Care Professional

**ICF** Informed Consent Form

**IRB** Institutional Review Board

LAR Legally Authorized Representative

NICU Neonatal Intensive Care Unit

PI Principal Investigator

**POC** Point Of Care

**SAE** Serious Adverse Event

**SADE** Serious Adverse Device Effect

**SCN** Special Care Nurseries

**SIV** Site Initiation Visit

UG User Guide

# 1.0 Identification of the Protocol/ Clinical Investigation Plan (CIP)

**1.1 Title of the clinical investigation**: Evaluation of the Performance of CONTOUR NEXT® and CONTOUR PLUS ELITE® Blood Glucose Monitoring Systems in Neonates using Capillary Blood Samples

**1.2 Protocol Number:** GCA-PRO-2021-003-01

**1.3 Date:** October 14, 2022

**1.4** Revision Status

| Date | Revision History |
|---|---|
| 30Jun2022 | Initial Release version |
| 14Oct2022 | 1. Amendment 1 |
| | Sections 3.0, 8.2, and 10.1.1: Changed "up to 150 subjects may be enrolled to obtain the required number of samples" to "up to 200 subjects may be enrolled to obtain the required number of samples." |
| | Section 13.1.2: Changed "meter results will be $2*120 = 240$ " to "meter results will be at least $2*120 = 240$ ." |
| | Section 13.10: Added "or valid" to the following statements: "Samples with no associated or valid hematocrit value." "Samples with no associated or valid Cobas 6000 value." |
| | Appendix D: Added "Ensure the tube setting on the HemataStat II™ is set to 0.5 mm ID (inner diameter)." |

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1

Ascensia Diabetes Care

Version: 14Oct2022


#### 2.0 Contact Information

**2.1** Sponsor: Ascensia Diabetes Care

100 Summit Lake Drive Valhalla, NY, 10595

Clinical Trial Manager contact:



**2.2** Principal Investigator (PI): Dennis Dietzen, PhD

2.2.1 Name, address, emergency contact details: St. Louis Children's Hospital

1 Children's Place

St. Louis, MO 63110

2.2.2 Professional position, roles, responsibilities and qualifications:

Professor of Pathology & Immunology, and Pediatrics, Washington University Medical Director, Laboratory Services, St. Louis Children's Hospital Medical Director, Laboratory Services, Children's Specialty Care Center, St. Louis PhD, Biochemistry and Molecular Biology, Indiana University School of Medicine

**2.3** Name and address of the investigation site: Site address is the same as in 2.2.1.

Business address of the site: Washington University

One Brookings Drive Campus Box 1054 St. Louis, MO 63130

- **2.4** Name(s) and address(es) of other institutions involved: Not Applicable
- **2.5** Description of study financing and the agreement between the sponsor/site.

Separate document: Clinical Trial Agreement between Ascensia Diabetes Care and Washington University, St. Louis.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1 Version: 14Oct2022

# 3.0 Synopsis of the Clinical Study

| Design Type: | Open Label, prospective, single arm study |
|---|---|
| Investigational Devices: | CONTOUR NEXT ® Blood Glucose Monitoring System (BGMS) |
| | CONTOUR PLUS ELITE® Blood Glucose Monitoring System |
| Trial objective | The purpose of this study is to extend the intended use of two BGMSs to include testing of neonatal blood by Health Care Professionals in a clinical setting for the quantitative measurement of glucose levels in neonates. |
| | This trial will evaluate the performance of both the CONTOUR NEXT BGMS and CONTOUR PLUS ELITE BGMS using blood from neonates within a hospital ward, e.g. routine/newborn nurseries, Special Care Nurseries, Neonatal Intensive Care Unit (NICU). The investigational BGMSs will be tested by a Point-of-Care operator using residual heel-stick capillary blood samples from neonates who underwent routine prescribed testing. |
| Reference Analyzer | Cobas® 6000 |
| Sample size: | A total of 120 blood samples tested in duplicate with N=240 evaluable results are required for this study. Therefore, at least 120 subjects will be enrolled. Up to 200 subjects may be enrolled to obtain the required number of samples. |
| | A sub-group of at least 5 capillary whole blood samples will be tested in neonates who are less than 24 hours of age. A sub-group of at least 5 capillary whole blood samples will be tested in neonates from the NICU. |
| Inclusion and <u>Inc</u> | clusion Criteria |
| Exclusion • | Residual capillary (heel-stick) blood samples collected from neonates (less |
| criteria: | than 28 days of age) after birth as part of prescribed testing. |
| • | Sample blood volume must be sufficient to complete investigational testing |
| | in addition to routine prescribed clinical laboratory testing. |
| Ex | clusion Criteria |
| • | Samples from subjects who are $\geq 28$ days of age. |
| • | Samples from subjects who have previously been enrolled into this study. |

Ascensia Diabetes Care


| Objectives The primary objective of the study is to evaluate the performance of and NEXT and CONTOUR PLUS ELITE BGMSs with residual neo samples. The performance of the BGMSs will be analyzed accordiologing objectives: | |
|---|---|
| Primary Objective: | |
| • At least 95% of all blood glucose results shall fall within ±12.5% of reference values (laboratory method) for glucose concentration ≥100 mg/dL mmol/L) and within ±12 mg/dL (±0.67 mmol/L) at glucose concentration <100 mg/dL (5.55 mmol/L). | |
| | • At least 98% of values shall be within ±20% of reference values (laboratory method) for glucose concentration ≥75 mg/dL (4.16 mmol/L) and within ±15 mg/dL(±0.83 mmol/L) at glucose concentrations < 75 mg/dL (4.16 mmol/L). |
| Number of stud | dy sites 1 site |
| Proposed start | date July 2022 |
| Study Duration | The study duration is expected to be approximately 4 months. The duration of each subject's participation is not applicable because the study uses residual samples. |

# 4.0 Identification and description of the investigational device

#### 4.1 Name of the investigational device:

- CONTOUR NEXT blood glucose monitoring system (Meter, CONTOUR NEXT Test Strips, Control solutions)
- CONTOUR PLUS ELITE blood glucose monitoring system (Meter, CONTOUR PLUS Test Strips, Control solutions)

# 4.2 <u>Intended purpose of investigational devices</u>

4.2.1 The CONTOUR NEXT and CONTOUR PLUS ELITE blood glucose monitoring systems (BGMS) are investigational BGMSs comprised of the blood glucose meter, the compatible test strips, and control solutions. They are automated systems intended for the quantitative measurement of glucose in fresh capillary whole blood drawn from the fingertip or palm, arterial blood, and venous blood. Its use in this trial is for the quantitative measurement of glucose levels in neonates from fresh capillary whole blood drawn from the heel.

Ascensia Diabetes Care


4.2.2 The system is intended to be used for self-testing by lay persons with diabetes and for near-patient testing by Health Care Professionals (HCP) to monitor the effectiveness of diabetes control.

- 4.2.3 The BGMS can only be used for monitoring blood glucose levels and is not for diagnosis or screening of diabetes. The system is intended for *in vitro* diagnostic use only.
- **4.3** Ascensia Diabetes Care (ADC) is the manufacturer of the device.
- **4.4** Traceability of the devices is achieved by serial numbers on the meters and lot numbers of the test strips and controls.
- **4.5** The population for which the device is intended in this study is residual blood sampled from neonates in a hospital setting.
- **4.6** No contact between the devices and the patients is required since all testing will be performed on blood sampled from a tube.
- **4.7** The technical and functional features of the investigational devices, CONTOUR NEXT and CONTOUR PLUS ELITE BGMSs, can be found in the User Guides (UG) in Attachments 1 and 2.
- **4.8** The instructions for use for the devices are found in the UGs (Attachments 1 and 2).
- **4.9** Training and experience required for use of the device is Good Clinical Practice (GCP) training, and laboratory experience. The study staff will be provided specific device training as part of the Site Initiation Visit (SIV) by the sponsor.

# 5.0 Justification for the Design of the Clinical Study

Hypoglycemia is the most common metabolic disturbance occurring in the neonatal period, which can lead to neonatal morbidity and developmental sequelae. Screening at-risk infants and the management of low blood glucose levels in the first hours to days of life is a frequent issue in the care of newborn infant. Transitional neonatal hypoglycemia usually resolves within 2 or 3 days of age. Severe prolonged neonatal hypoglycemia can cause seizures, brain damage, and neurodevelopmental impairment. Signs of neonatal hypoglycemia are non-specific, and babies with hypoglycemia are frequently asymptomatic. Therefore, it is common to screen babies considered at high risk for neonatal hypoglycemia with repeated blood glucose measurements. Usually, plasma or serum samples are used for routine blood glucose estimation in a hospital laboratory. However, such an approach using a laboratory-based testing method is not practical in acute situations due to the delayed turnaround time. Therefore, BGMS are frequently used for the bedside estimation of blood glucose levels. Rapid measurement time, smaller volume of required blood samples, and enhanced usability are the main benefits of using BGMS compared with laboratory-based testing. Most BGMS that are currently used are initially developed for monitoring blood glucose levels in adult patients with diabetes. Neonatal blood differs from adult blood in two major aspects—it has lower concentrations of blood glucose and a wider range of hematocrit levels (Adamkin 2011; BAPM 2017; Harris et al 2012; Lucas et al 1988; Movalia and Ogino 2006; Nuntnarumit et al 2011; Roth-Kleiner et al 2010; Rozance 2006).

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1


The CONTOUR NEXT and CONTOUR PLUS ELITE BGMSs are investigational BGMSs comprised of the blood glucose meter, the compatible test strips, and control solutions. They are automated systems intended for the quantitative measurement of glucose in neonatal blood, venous blood, fresh capillary whole blood drawn from the fingertip or palm. The system is intended to be used for self-testing by lay persons with diabetes and for near-patient testing by HCPs to monitor the effectiveness of diabetes control. Its use in this trial is for the quantitative measurement of glucose levels in neonates from fresh capillary whole blood drawn from the heel by HCPs in a clinical setting.

This investigational clinical trial will evaluate the performance of two BGMSs, CONTOUR NEXT BGMS and CONTOUR PLUS ELITE BGMSs, in neonates within a hospital ward, e.g. routine/newborn nurseries, Special Care Nurseries (SCN), Neonatal Intensive Care Units (NICU). The BGMS will be used by a POC operator in a clinical setting using residual heel-stick capillary blood samples from neonates who underwent routine prescribed testing. The residual blood no longer needed for clinical purposes will be used for this study.

#### 6.0 Risks and benefits of the investigational device and clinical investigation

#### Risks

This is a low risk study. Residual blood samples will ONLY be tested for the study if the neonate is having prescribed blood tests done as ordered by their physician. Therefore, there will be no additional blood samples collected for this study. All testing procedures with the investigational device will be performed by the study staff in a laboratory setting and at no point will the neonate come in contact with the Investigational device or any other study-related material. There is no discomfort to the neonate as only residual blood will be collected.

There are no risks to patients associated with this study except for the potential for loss of confidentiality. Measures will be taken to minimize this risk by de-identifying study samples. Without the identification list that is exclusively stored at the site, connection between personal data and study data is not possible.

#### Benefits

There are no direct benefits to the subject (neonate) for donation of residual blood samples for this study except to contribute to a study that provides information on the performance of two BGMSs when measuring glucose in capillary blood by HCPs within a clinical setting. Subjects will not receive compensation.

There are no anticipated adverse device effects.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1 Ascensia Diabetes Care CONFIDENTIAL

# 7.0 Objectives and Hypotheses


The primary objective of the study is to evaluate the performance of CONTOUR NEXT and CONTOUR PLUS ELITE BGMSs with residual heel-stick capillary blood samples from neonates, i.e. babies who are less than 28 days old. The performance of the BGMS will be analyzed according to the following objectives:

- 7.1 **Primary Objective**: The accuracy criteria below are taken from CLSI. *Point-of-Care Blood* Glucose Testing in Acute and Chronic Care Facilities; Approved Guideline – Third Edition. CLSI document POCT12-A3. Wayne, PA: Clinical and Laboratory Standards Institute; 2013.
  - At least 95% of all blood glucose results shall fall within ±12.5% of reference values 7.1.1 (laboratory method) for glucose concentration ≥100 mg/dL (5.55 mmol/L) and within  $\pm 12 \text{ mg/dL}$  ( $\pm 0.67 \text{ mmol/L}$ ) at glucose concentrations <100 mg/dL (5.55 mmol/L).
    - Note: Satisfying Criterion 7.1.1 would also satisfy the ISO 15917:2013 criteria of obtaining the  $\pm 15\%$  of reference values (laboratory method) for glucose concentration  $\geq 100 \text{ mg/dL}$  (5.55 mmol/L) and within  $\pm 15 \text{ mg/dL}$  ( $\pm 0.83 \text{ mmol/L}$ ) at glucose concentrations <100 mg/dL (5.55 mmol/L).
  - 7.1.2 At least 98% of values shall be within  $\pm 20\%$  of reference values (laboratory method) for glucose concentration  $\geq$ 75 mg/dL (4.16 mmol/L) and within  $\pm$ 15 mg/dL ( $\pm$ 0.83 mmol/L) at glucose concentrations < 75 mg/dL (4.16 mmol/L).

#### Other Objectives: 7.2

- Evaluate the performance of both BGMSs for neonates who are <24 hours old. Compute differences between BGMS and laboratory blood glucose measurements and plot them against hematocrit results.
- Evaluate the performance of both BGMSs with blood samples from babies in the NICU.
- Compute differences between BGMS and laboratory blood glucose measurements and plot them against bilirubin results, for those subjects where bilirubin measurements were recorded (when available).

# 8.0 Clinical Study Design

- 8.1 This is an open label, prospective, single arm study. The results of the study devices will be compared to the laboratory analyzer results from the same blood sample.
- For each BGMS, 120 evaluable samples (N=240 evaluable results due to duplicate testing) 8.2 are required. Therefore at least 120 subjects will be enrolled. Up to 200 subjects may be enrolled to obtain the required number of samples.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1

Ascensia Diabetes Care

Version: 14Oct2022


#### 8.3 Randomization:

- 8.3.1 Since two BGMSs will be tested in the study, the order of testing the study devices will be randomized.
- 8.3.2 Three strip lots (per BGMS) will be tested, with each sample tested with one lot. The strip lots will be randomized.
- **8.4** The results from these two BGMSs will not be compared to each other.
- **8.5** The study design follows CLSI- POCT12-A3:2013 and ISO 20916:2019(E) to ensure it is scientifically robust and valid.
- 8.6 Subjects with non-evaluable data will be replaced as needed to obtain N=120 samples, and N= 240 results (duplicate results) for each BGMS.

#### 9.0 Investigational device(s) and comparator(s)

#### 9.1 Materials and Methods

- 9.1.1 Resources Supplied by Investigator Staffing
- Principal Investigator / and, if applicable, Sub-Investigators
- HCP to collect blood samples
- Laboratory professionals to perform meter testing, hematocrit, and laboratory analyzer testing
  - 9.1.2 Resources Supplied by Investigator Other
- Hospital IRB and/or Central IRB approval of the protocol.
- Facility with adequate laboratory resources for conducting all tests (including blood glucose laboratory analyzer, hematocrit measurement instrument).
- Facility with adequate neonatal population for at least 120 study-appropriate samples within the desired course of the trial.
- Cobas<sup>®</sup> 6000 (Roche Diagnostics Corp., Indianapolis, IN) Laboratory Analyzer, to measure glucose in plasma.
- Print-outs of the Cobas 6000 results for Quality Control (QC) checks during study days.
  - 9.1.3 Resources Supplied by Ascensia Materials
  - Protocol and sample Case Report Forms (CRF)
  - CONTOUR NEXT® meters
  - CONTOUR NEXT® strips (3 lots) with inserts
  - CONTOUR NEXT® UGs

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1 Ascensia Diabetes Care CONFIDENTIAL

- CONTOUR PLUS ELITE® meters
- CONTOUR PLUS® strips (3 lots) with inserts
- CONTOUR PLUS ELITE® UGs
- CONTOUR NEXT® and CONTOUR PLUS® Low, Normal and High Control solutions with inserts
- Hematocrit instrument and testing supplies
- Thermometer/hygrometers for measuring environmental conditions at the meter testing location, if needed. The site may use its calibrated measuring devices with approval of ADC.
- Disinfectant (see Appendix A for procedure and detail)
- Serum controls for the laboratory glucose analyzer
- Atomic clock(s)
- 9.2 Note that the subjects will not be exposed to the study devices since residual blood samples will be collected in a tube and used for all study procedures.
- All meters will have Bluetooth® ON. 9.3
- The meters, test strips, and CONTOUR NEXT and PLUS control solutions must be stored 9.4 at 9-30C. See Appendix C for serum control storage.

# 10.0 Subjects


#### 10.1 Recruitment and Enrollment

- 10.1.1 A total of at least 120 blood samples with evaluable results (N=240) are required for this study. Up to 200 subjects may be enrolled into the study to obtain the required number of samples. See section 13.10 for the definition of evaluability.
- 10.1.2 The subject population will consist of neonates from hospital wards (e.g. routine/newborn nurseries, SCN, NICU) of the clinical investigational site.
- 10.1.3 There will be a sub-group of at least 5 samples collected from neonates who are less than 24 hours of age.
- 10.1.4 There will be a sub-group of at least 5 samples collected from neonates from the NICU.
- 10.1.5 The samples in these two sub-groups are permitted to overlap.
- 10.1.6 The study staff will document subject demographics, including age and gender.

Ascensia Diabetes Care


10.1.7 Unused residual blood samples collected for study testing procedures will be discarded according to hospital Laboratory Safety Guidance (Occupational Safety and Health Administration) procedures.

#### 10.2 <u>Inclusion Criteria</u>

- 10.2.1 Residual capillary (heel-stick) blood samples from neonates (less than 28 days of age) after birth as part of prescribed testing.
- 10.2.2 Sample blood volume must be sufficient to complete investigational testing in addition to routine prescribed clinical laboratory testing.

#### 10.3 Exclusion Criteria

- 10.3.1 Samples from subjects who are  $\geq$  28 days of age.
- 10.3.2 Samples from subjects who have previously been enrolled into this study.

## 10.4 Study Duration

- 10.4.1 The total expected duration to complete the clinical investigation is ~4 months.
- 10.4.2 The expected duration of each subject's participation is not applicable since there is no direct subject participation. Only residual blood samples from subjects will be tested per the study procedures only on the day of sample collection.

#### 11.0 Procedures

#### 11.1 Summary

Laboratory professionals will test the glucose concentration of residual capillary whole blood samples, collected (into a tube) from neonatal heel-sticks only, using the CONTOUR NEXT and CONTOUR PLUS ELITE BGMSs. The investigational site will enroll neonates from hospital wards (e,g, routine/newborn nurseries, SCN, NICU). For subject safety and ethical reasons, only those neonates already scheduled to have blood samples obtained for prescribed testing (by the hospital staff), will be enrolled into this study. No neonate will have heel-stick blood collected solely for the purpose of this study.

A minimum of 10 capillary whole blood samples (from residual neonatal heel-stick) will be tested in duplicate on both BGMSs. A sub-group of at least 5 of these blood samples will be from neonates who are less than 24 hours of age. A sub-group of at least 5 blood samples will be from neonates in the NICU. These two sub-groups' samples are permitted to overlap.

Up to 50uL of whole blood will be removed from the subject's sample tube, and will be used for completing a total of 4 tests using both BGMSs (two tests with CONTOUR NEXT BGMS and two tests with CONTOUR PLUS ELITE BGMS), and a hematocrit measurement. Each subject sample will be tested using both BGMS as per the randomization schedule. After completion of the BGMS testing, each meter will be cleaned and disinfected as per the procedures in Appendix A.


The site staff will use their Laboratory Glucose Analyzer (approved by the Sponsor) for the laboratory assessment of blood glucose samples tested in duplicate as part of prescribed testing of the same sample. The laboratory duplicate results will be averaged. In cases where the prescribed test for the sample is a bilirubin analysis, the results of this test will be recorded as part of the study data.

During the study, three test strip lots will be used for each BGMS. The test strip lots will be arbitrarily designated as green, blue, or red to easily identify the bottles during the study. See Table 1 for the description of test strip distribution during the study. Blood samples will be assigned to one of three test strip lots. The assignment will be made in a rotating order following the random order in which samples are received. For each sample, the order of testing each of the two BGMSs will also be randomized.

Meter System & **Green Lot** Red Lot **Blue Lot** Test Strips CONTOUR NEXT Meter 40 Samples 40 Samples 40 Samples (CONTOUR NEXT Test Strips) ~80 tests ~80 tests ~80 tests CONTOUR PLUS ELITE Meter 40 Samples 40 Samples 40 Samples (CONTOUR PLUS Test Strips) ~80 tests ~80 tests ~80 tests

Table 1. Strip Lot Assignments Per Meter Type

# 11.2 Study Staff Training

The site study staff will be given copies of the protocol and meter instructional material (UG). They will participate in a training session conducted by the Ascensia Study team or designee. The training will be documented, and the following will be reviewed:

- 11.2.1 Protocol & CRFs
- 11.2.2 Meter Instructions for Use (UG)
- 11.2.3 Meter control solution testing
- 11.2.4 Error messages and troubleshooting
- 11.2.5 GCP
- 11.2.6 Practice using the CONTOUR NEXT and CONTOUR PLUS ELITE BGMSs
- 11.2.7 Practice preparing and reading hematocrit samples

#### 11.3 Meter Control Solution Testing

Control testing on the study BGMS will occur after they arrive at the site and before the trial starts.

Ascensia Diabetes Care


11.3.1 The site staff will equally distribute (approximately) the strip lots for control testing.

- 11.3.2 The site staff will perform 3 control tests (one each of low, normal, and high) on each BGMS assigned for the study.
- 11.3.3 Results will be recorded and compared to the control ranges listed on the test strip bottle.
- 11.3.4 If results are out of range, troubleshooting will be performed (see UG), and the test will be repeated for a total of up to 3 attempts.
- 11.3.5 If the meter tests are out of range after troubleshooting is complete, the meter will be removed from the study, and the Ascensia Study Manager will be notified. Additionally, this will be documented on the 'Device Deficiency Reporting Form'.

#### 11.4 Blood Glucose Testing

- 11.4.1 No blood will be taken from study subjects solely for this study. Neonatal blood will be collected for prescribed testing and residual blood from the sample will be used for this study. Blood will be collected following HCP's orders by nursing/phlebotomy staff using standard heel puncture techniques. All samples will be transported to the laboratory per standard practice and submitted for prescribed clinical testing. Samples will be collected according to hospital standards and procedures and will be collected into a tube containing anticoagulants (lithium heparin).
- 11.4.2 Neonatal blood samples will be inspected to verify if the volume drawn was sufficient to complete both prescribed clinical and investigational testing by laboratory personnel. Samples that do not have sufficient volume to complete the required investigational testing will not be used for the clinical trial.
- 11.4.3 If sufficient volume is available, this is the time of enrollment. No more than the agreed amount (50 uL) of capillary whole blood will be removed from the original sample to perform blood glucose testing on two investigational BGMSsand a hematocrit measurement.
- 11.4.4 The collected samples will be used within a maximum of 5 h of sample collection time, and will be kept at room temperature (23  $\pm$  5 °C) before evaluation.
- 11.4.5 Each blood sample for the study will be assigned an ID that is not traceable to the identity of the subject. The first digit will indicate the site ID followed by three digits indicating the sample ID as follows: X-001, X-002, X-003, and so on.
- 11.4.6 Strip lot (color code) will be determined via a randomization schedule provided by the Sponsor. The testing order of the meter will also be based on a randomization schedule. Note that one CONTOUR NEXT and one CONTOUR PLUS ELITE BGMS per subject will be used and the meters will be disinfected after use as per procedures listed in Appendix A.

11.4.7 For each subject, a CONTOUR NEXT BGMS, and a CONTOUR PLUS ELITE BGMS will be brought to the testing area. A test strip (as assigned for the given BGMS) will be inserted into each of the 2 meters (same color code strip lot for both meters).

- 11.4.8 A drop of blood will be placed on a piece of Parafilm (or other non-absorbent material) and immediately tested with the first and second meter.
- 11.4.9 The test strips in the two meters will then be replaced, to prepare the meters for duplicate testing.
- 11.4.10 A new drop of blood will be placed on the Parafilm and immediately tested with the first and second meter.
- 11.4.11 A hematocrit measurement (%) will also be performed. (See Section 11.6.)
- 11.4.12 The blood (from the same sample as used in meter testing) will be centrifuged within 10 minutes of BG testing for separation into plasma.
- 11.4.13 The start time of centrifugation will be recorded. Centrifugation must be performed within 10 minutes of the first-meter assay.
- 11.4.14 The plasma will be tested in duplicate with the laboratory analyzer within 60 minutes of the meter test. If greater than 60 minutes of the meter test, plasma samples may be refrigerated.

#### **11.5 Errors**

- 11.5.1 If the meter reports an error code during blood glucose testing, the instructions shown in the UG should be followed. Re-testing is recommended (per the UG). The reason for the repeated test will be documented in the comments section of the form. No more than a total of 3 attempts are allowed.
- 11.5.2 The study staff will record all meter error codes as appropriate for the meter tests as it occurs.

#### 11.6 Hematocrit

- 11.6.1 At least one hematocrit tube, but preferably two, will be filled with the residual whole blood and then centrifuged.
- 11.6.2 The hematocrit will be measured from only one tube; the second tube will be collected as a backup in case the first tube is not measurable (i.e., tube spun out, broken tube, clay seal compromised, etc.). Additional details regarding hematocrit measurements are found in Appendix D.

#### 11.7 Testing Schematic

**Table 2. Sample Testing Schematic** 

| Step | Test/action | Description |
|---|---|---|
| 1 | Sample prep | <ul> <li>Ensure collection of residual neonatal sample in collection tube containing anticogulant (lithium/heparin).</li> <li>Confirm sufficient blood volume to perform all testing procedures.</li> <li>If so, then aliquot up to 50 uL into microtube and cover.</li> </ul> |
| 2 | Testing prep | Assign one CONTOUR NEXT meter and one CONTOUR PLUS ELITE meter to the patient sample. Follow the strip lot randomization (red, green, blue) and get the test strip bottle for the respective meter. Get a piece of parafilm. For steps 3 and 4, follow meter test order per randomization schedule. |
| 3 | Meter Test 1 | <ul> <li>Put a test strip into each meter.</li> <li>Immediately place 1 drop of blood on the parafilm and test with both meters. Record results.</li> <li>In case of error, may repeat 2 more times with a new blood drop.</li> <li>Record time of successful meter tests.</li> </ul> |
| 4 | Meter Test 2 | Replace test strips, and place new blood drop on parafilm to repeat Step 3 for duplicate testing. |
| 5 | Hematocrit | <ul> <li>Using the blood from the same collection tube, fill up to 2 hematocrit tubes.</li> <li>Perform hematocrit measurement, and record results.</li> </ul> |
| 6 | Centrifugation | ■ Centrifuge blood, and record start time. (The centrifugation start time must be within 10 min of meter tests). |
| 7 | Laboratory tests* | <ul> <li>Perform blood glucose testing of plasma sample on laboratory analyzer (Cobas) in duplicate.</li> <li>Record results.</li> </ul> |

<sup>\*</sup> Pre-study and on-study serum control testing on Cobas: See 11.8 and Appendix C.

#### 11.8 Accuracy and Precision of Cobas 6000

Performance of the Cobas 6000 will be tracked by two methods. The primary method will be the instrument QC check procedure regularly applied by the clinical site. In addition, serum controls will be provided by Ascensia for internal research purposes only, and will not impact the study data or data collection. See Appendix C for further details.

#### 11.9 Bilirubin Data

Bilirubin data will be collected to assess potential interference with elevated bilirubin levels occurring in neonates. In cases where the prescribed test for the sample is a bilirubin analysis, the results of this test will be recorded as part of the study data from the hospital records.

No bilirubin test will be performed on study samples just for the purpose of this study. Thus, not all study samples may have bilirubin data.

#### 11.10 Temperature and Humidity Logs

• The study staff will measure the temperature/humidity in the meter testing area once during the day that meter testing occurs and record the results on the appropriate log form.

• Study staff will maintain a temperature log for the storage of investigational materials including the meters, test strips, controls, and serum controls.

# 12.0 Monitoring Plan

- **12.1** A monitoring plan will be completed by the Study Manager/designee prior to the study.
- **12.2** The study manager or designee will conduct the SIV. The frequency of the number of monitoring visits by sponsor personnel or designee(s) will be based on the monitoring plan and will include at least 1-3 monitoring visits and a close-out visit.
- **12.3** Sponsor representatives may observe some study testing as part of study monitoring. This will be done under supervision of the Investigator.
- **12.4** Sponsor representatives will maintain subject confidentiality, and will not interfere with the rights of human subjects or safety, or bias study conduct.

#### 13.0 Statistical Plan

#### 13.1 <u>Sample Size</u>

- 13.1.1 The sample size requirement is based on the primary objective, section 7.0.
- 13.1.2 There will be a minimum of N = 120 study samples entered into the study. The meter results will be taken in duplicate, so that the total sample size of meter results will be at least 2\*120 = 240.
- 13.1.3 With a sample size of n = 240 results, there is approximately a 95% chance that at least 228 of those results (95% of 240) will be "accurate" (errors within either  $\pm 12$  mg/dL ( $\pm 0.67$  mmol/L) when the comparator result is < 100 mg/dL (5.55 mmol/L), or  $\pm 12.5\%$  when the comparator result is  $\geq 100$  mg/dL (5.55 mmol/L) if the evaluation (meter) system has a 96.77% chance of yielding an "accurate" result.
- 13.1.4 Conversely, there is about a 95% chance of obtaining fewer than 228 "accurate" results if the system only has an approximately 92.03% chance of yielding an accurate result.
- 13.1.5 Note that each glucose result obtained with the evaluation devices will be considered either 'accurate' or 'not accurate', where accuracy depends on the particular test criterion as described in section 7.0 of this protocol.


#### **13.2 Blood Glucose Measurements**

Data analysis follows analyses and presentations described in CLSI. *Point-of-Care Blood Glucose Testing in Acute and Chronic Care Facilities; Approved Guideline – Third Edition*. CLSI document POCT12-A3. Wayne, PA: Clinical and Laboratory Standards Institute; 2013.

The unit conversion formula for blood glucose is the following:

Xmmol/L = Ymg/dL / 18.016

#### 13.3 Bland-Altman Plots

Modified Bland-Altman plots (the difference between each evaluation device results and reference results plotted against reference results) will be constructed.

#### 13.4 Weighted Least Squares Regression

Weighted least squares regressions of meter results against comparator results will be performed. If *M* represents the meter result, and *C* the comparator result, the linear model can be expressed as:

$$M = \beta_0 + \beta_1 C + \varepsilon$$
$$\varepsilon \sim N(0, cv * C)$$

The parameter *cv* is the coefficient of variation, which is assumed to be constant across the glucose range. The weighting function will be:

$$w = C^{-2}$$

This weighting function is used to account for the constant cv nature of glucose measurement (Draper and Smith, 1998).

#### **13.5** Accuracy Analyses

13.5.1 Two sets of metrics will be calculated:

Relative (Percent) Difference (RD) for reference result  $\geq$  threshold glucose:

$$RD = \frac{M-C}{C} 100\%$$

where: M = strip/meter result and C = comparator or reference method result.

Difference (D) for reference result < threshold glucose:

$$D = M - C$$


#### 13.5.2 Primary objective:

The threshold glucose value is 100 mg/dL (5.55 mmol/L). Accuracy will be assessed using the CLSI. *Point-of-Care Blood Glucose Testing in Acute and Chronic Care Facilities; Approved Guideline – Third Edition*. CLSI document POCT12-A3. Wayne, PA: Clinical and Laboratory Standards Institute; 2013.

i.e., D within  $\pm 12 \text{ mg/dL} (\pm 0.67 \text{ mmol/L})$  for comparator result < 100 mg/dL (5.55 mmol/L) and RD within  $\pm 12.5\%$  for comparator result  $\ge 100 \text{ mg/dL} (5.55 \text{ mmol/L})$ .

For RD, the percent of results within  $\pm 5\%$ ,  $\pm 10\%$ ,  $\pm 12.5\%$ ,  $\pm 15\%$  and  $\pm 20\%$  will be computed.

For D, the percent less than or equal to  $\pm 5$  mg/dL ( $\pm 0.28$ mmol/L),  $\pm 10$  mg/dL ( $\pm 0.56$  mmol/L),  $\pm 12.0$  mg/dL ( $\pm 0.67$  mmol/L),  $\pm 15$  mg/dL ( $\pm 0.83$  mmol/L), and  $\pm 20$  mg/dL ( $\pm 1.11$  mmol/L) will be computed.

The *RD* and *D* distribution tables will be constructed using a threshold of 100 mg/dL(5.55 mmol/L).

As discussed in section 13.1 (Sample Size), with n = 240, the critical number (minimum) of accurate results is 228, which yields approximately 95% chance of satisfying the criterion if the actual probability that any result will be accurate is at least 96.77%. Symbolically, this criterion is equivalent to testing the hypothesis:

 $H_0: Prob\{accurate\} < 96.77\%$  versus the alternative:

 $H_1: Prob{accurate} \ge 96.77\%$ 

This test has a power of about 95%, with n =240, to reject  $H_0$  if the actual probability of obtaining an accurate result is 96.77%. Conversely, there is about a 95% chance that the null will NOT be rejected if the actual probability that a result with the evaluation device would satisfy this definition of accuracy is only about 92.03%.

#### 13.5.3 The second part of the primary objective

The second part of the primary objective states that at least 98% of the n = 240 results must fall within  $\pm 15$  mg/dL( $\pm 0.83$  mmol/L) of the comparator result (comparator < 75 mg/dL/4.16 mmol/L)) or  $\pm 20\%$  of the comparator result (comparator  $\geq 75$  mg/dL/4.16 mmol/L). Thus, with n = 240, there must be at least 236 BGMS results satisfying this requirement. This is equivalent to testing the hypotheses:

*H*<sub>0</sub>:  $Prob\{accurate\} < 98.33\%$  versus the alternative:

 $H_1$ :  $Prob{accurate} \ge 98.33\%$ 

There is approximately a 95% chance of rejecting  $H_0$  in favor of  $H_1$  if the actual probability that a meter measurement would satisfy the  $\pm 15$ mg/dL or 20% is 98.33%. Conversely, there is about a 95% chance that the null will NOT be rejected if the actual probability that a result with the evaluation device would satisfy this definition of accuracy is only about 96.23%. It is possible

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1 Ascensia Diabetes Care CONFIDENTIAL

that the sample size after the study is completed may not be exactly 240. The critical values will be approximately 95% or 98% of results (first and second parts of primary objective, respectively), and the associated hypotheses will be adjusted to reflect the change while maintaining no more than a 95% chance of rejecting the null hypotheses.

#### 13.6 Neonates < 24 hrs. old and Neonates in NICU – Other Objectives

In addition to the neonates less than 28 days of age, additional analyses of data from neonatal subjects ≤ 24 hrs. old and neonates in NICU will be performed.

- 13.6.1 Specifically, differences in BG results between BGMS and reference laboratory instrument will be plotted against the laboratory instrument results (modified Bland-Altman plot).
- 13.6.2 There must be at least 5 subjects <24 hrs. old and 5 subjects in NICU enrolled to perform this analysis. These groups may have any or all subjects in common.

#### **13.7** <u>Hematocrit Analysis – Other Objectives</u>


- 13.7.1 Hematocrit will be measured for each subject. Mean, median, minimum, maximum, and standard deviation, will be computed for hematocrit determinations.
- 13.7.2 The effect of hematocrit on meter results will be presented via regression of differences between the meter and laboratory BG measurements against hematocrit.

#### **13.8** <u>Bilirubin Analysis – Other Objectives</u>

For neonates who would have bilirubin results, regression analysis will be used to assess the effects of bilirubin on the difference between meter and laboratory reference method blood glucose measurements.

There must be at least 3 subjects enrolled with bilirubin recorded to perform this analysis. If fewer than 3, then the results will be reported in a table.

#### **13.9** Temperature and Humidity

Mean, median, standard deviation, minimum and maximum room temperature, and humidity will be computed.

#### 13.10 Data Evaluability

Blood glucose data will be considered not evaluable for the following reasons:

- Samples with no associated or valid hematocrit value.
- Samples with no associated or valid Cobas 6000 value.

• Failure to begin to separate the plasma from the red cells within 10 minutes of obtaining the first meter test.

- The collected samples exceed a maximum of 5 h of sample withdrawal time, and will be kept at room temperature  $(23 \pm 5 \, ^{\circ}\text{C})$  before evaluation.
- For a given sample, the meter is missing a replicate.
- Results of the glucose analyzer blood sample are not within ±4% of each other, 100\* (Rep2-Rep1)/Rep1, or ±4mg/dL (0.22mmol/L) of each other (Rep2-Rep1) if the average falls below 100mg/dL (5.5mmol/L).

# 14.0 Data Management

- **14.1** A unique number will identify each subject/sample. The unique number will be entered on the CRFs. The site will create a procedure to de-identify subjects from samples so that the staff members documenting subject names will not have access to sample results and the staff members testing the samples will not have access to subject names. A master list of subject names, with their subject IDs, will be kept by the Investigator at the study site until the study has been closed.
- **14.2** Study personnel will complete and sign all appropriate forms in compliance with GCP. CRFs should be completed legibly, in black or blue ink. If it is necessary to make corrections, a single line should be drawn through the original entry, the new entry is written in, and the correction initialed and dated by the individual correcting the CRF.
- **14.3** Study data will be primarily collected through an electronic data capture (EDC) system used by Ascensia. The data will be recorded on forms by designated study staff that will serve as source documents and entered into the EDC system. All source forms will be retained by the site.
- **14.4** In addition to data collection, the EDC system will be used for data cleaning as well as monitoring operations. Site users will be trained on this system before the start of the study and their access to EDC system will be contingent upon successful completion of training requirements.

#### 15.0 Amendments to the Protocol

- **15.1** Any change to this protocol requires a protocol amendment (or revision) unless the IRB agrees to an administrative change (for minor changes).
- **15.2** Determine the justification(s) for the protocol revision, impact of the changes on subject safety, the clinical or statistical significance of the data, impact of changes on the clinical investigators and their staff, and impact on timely completion of the clinical trial.
- **15.3** Determine if the revision meets the criteria of a Substantial Amendment.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1

Ascensia Diabetes Care Version: 140ct2022 CONFIDENTIAL

#### **15.4** Substantial Amendments

15.4.1 Substantial amendments to the conduct of the clinical trial may arise from changes to the protocol or from new information relating to the scientific documents in support of the trial. Substantial changes require notification to the overseeing IRB before implementation. For any questions on whether a change would be considered substantial, consult with the respective IRB.

- 15.4.2 Amendments to the trial are regarded as "substantial" where they are likely to have a significant impact on the:
  - Safety, health or rights or physical or mental integrity of the subjects,
  - Scientific value of the trial including robustness or reliability of the data generated by the study,
  - Conduct or management of the trial,
  - Quality or safety of any investigational product used in the trial.
- 15.4.3 An amendment is only to be regarded as "substantial" when one or more of the above criteria are met but the IRB may have additional requirements that shall be considered.
- 15.4.4 Examples of substantial amendments may include (but are not limited to):
  - New tests
  - Increase in the number of visits due to safety issues associated with the ongoing trial
  - Change of inclusion/exclusion criteria
  - Change in the number of participants
  - Updated PI
  - Informed Consent Form (ICF)
  - Updated investigator brochure with relevant safety information
  - Change in the management of the study
  - Temporary halt to the study or restart of the trial after a temporary halt
- **15.5** Once justified, the protocol changes can be drafted and the changes documented in the Revision History. The changes are to be incorporated directly into the body of the protocol document itself (revised protocol).
- **15.6** Once the drafted revision is approved internally and by the PI, it will be submitted to the IRB, where required. All subsequent, IRB-approved, revised protocols would be numbered sequentially.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1

Ascensia Diabetes Care

Version: 14Oct2022


**15.7** The amended protocol will be approved by the original approvers, including the sponsor representatives or designee and the PI.

**15.8** The sponsor must assure that each investigator (and his/her staff) is following the most recent IRB approved amendment or revised protocol as the study proceeds. The sponsor must ensure that the study monitors, investigator(s) and study staff have been trained with respect to any recent protocol amendments and revisions prior to implementation.

# 16.0 Deviations from the clinical protocol

- **16.1** A protocol deviation is any alteration or modification to the procedures described in the protocol. The investigator is not allowed to deviate from the protocol. The only exceptions to this are:
  - 16.1.1 The deviation is necessary to protect the subject's rights, safety and well-being, or the scientific integrity of the clinical investigation without prior approval of the sponsor and IRB.
  - 16.1.2 Prospective deviations that broaden the scope of the protocol (waivers of the protocol) are prohibited. Under emergency circumstances, these instances can proceed.
- **16.2** Procedures for recording, reporting and analyzing protocol deviations will include recording the deviation on a Protocol Deviation log form to be supplied by the Sponsor.

# 17.0 Device Accountability

- **17.1** Description of the procedures for the accountability of investigational devices as follows:
  - 17.1.1 Access to investigational devices shall be controlled and the investigational devices shall be used only in the clinical investigation and according to the protocol.
  - 17.1.2 The sponsor shall keep records to document the physical location of all investigational devices from shipment of investigational devices to the investigation sites until return or disposal.
  - 17.1.3 Accountability: The PI or a delegate shall keep records documenting the receipt, use, return and disposal of the investigational devices, (including unused, expired or malfunctioning devices), which shall include:
    - Date of receipt
    - Identification of each device (serial number of meter or strip lot)
    - The expiry date, if applicable
    - Date(s) of use
    - Subject number

• Date of return of unused, expired or malfunctioning investigational devices, if applicable

## 18.0 Regulatory

Ascensia (sponsor) has determined that according to IDE requirements of 21 CFR 812.2(c), this IVD study meets all conditions for IDE exemption and therefore submission of an IDE application to FDA is not required. Determination is based on the following:

The Contour Next and Contour Plus Elite Glucose Monitoring Systems (IVDs);

- are labeled in accordance with 21 CFR 809.10(c)
- are non-invasive
- do not require an invasive sampling procedure that presents significant risk
- do not by design or intention introduce energy into a subject
- are not used as a diagnostic procedure without confirmation of the diagnosis by another, medically established diagnostic product or procedure.

#### 18.1 IRB Approval

- 18.1.1 Before study initiation, an IRB must review this protocol, the ICF, and any other supporting study documents which impact subject safety. The IRB will determine if the Informed Consent is required according to local regulations and requirements or if consent is not required (ISO 20916:2019(E)).
- 18.1.2 The investigational site may not begin the study until the IRB has given its written and dated approval via a letter that identifies the version/date of the protocol and ICF, if applicable, or a notification that consent is not required.
- 18.1.3 A copy of the IRB approval letter must be provided to the Investigator and to sponsor prior to the SIV.

#### **18.2 Study Documentation Procedures**

- 18.2.1 The investigator will keep study records for a minimum of three years. Alternatively, other arrangements may be made with Ascensia for study document storage.
- 18.2.2 Study Investigational Devices will be labeled "For Investigational Use only. The performance characteristics of this product have not been established" for this study.
- 18.2.3 After study completion, all BGMSs will be disinfected before they are returned to Ascensia. A decontamination log will be completed for the used meters. The meters, unused strip vials, control solutions, and meter UGs will be accounted for at the site and returned to the Ascensia Study Manager upon completion of the trial.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1 Ascensia Diabetes Care CONFIDENTIAL

18.3 <u>Investigator's Report of Study Closure</u>


# 18.3.1 Sponsor representatives will notify the site that the study is closed. The study will be considered closed when the data has been locked for data analysis.

- 18.3.2 The Investigator or designee will submit a report summarizing subject disposition and other study details, as appropriate, to the Study Manager and the IRB. This report will be completed within 3 months of the study closure date.
- 18.3.3 In addition, the Study Manager, or designee, will report the completion of the study to the IRB within 6 months of study closure.

# 19.0 Statements of compliance

- **19.1** This clinical investigation will be conducted in compliance with applicable requirements:
  - 19.1.1 Protection of Human Subjects regulations in 21 CFR part 50.
  - 19.1.2 IRB regulations in 21 CFR part 56.
  - 19.1.3 Investigational Device Exemptions regulations in 21 CFR part 812.
  - 19.1.4 Declaration of Helsinki.
  - 19.1.5 CLSI. Point-of-Care Blood Glucose Testing in Acute and Chronic Care Facilities; Approved Guideline - Third Edition. CLSI document POCT12-A3. Wayne, PA: Clinical and Laboratory Standards Institute; 2013.
  - 19.1.6 International Standards: ISO20916:2019(E) In vitro diagnostic medical devices Clinical performance studies using specimens from human subjects – Good Study Practice and In Vitro Diagnostic Regulation 2017/746 Annex XIII, Part 2.
  - 19.1.7 British Standard BS EN 13612:2002, "Performance evaluation of in vitro diagnostic medical devices."
- **19.2** The clinical study shall not begin until the required approval from the IRB or regulatory authority have been obtained.
- **19.3** Clinical trial insurance shall be provided as appropriate.

#### **20.0 Informed Consent Process**

The IRB will determine if the Informed Consent is required according to local regulations and requirements for use of residual blood samples for this study.

The following will only apply if Informed Consent is required by the IRB. If the IRB determines that consent is not required, this section will not apply.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1 Ascensia Diabetes Care CONFIDENTIAL

20.1 Since the subject is a neonate, the subject's parent/guardian - Legally Authorized Representative (LAR) - will complete the informed consent process before performing any study procedures.

- 20.2 The LAR will be informed about the study objectives, investigational devices, study procedures, expected study duration, and risks of study participation.
- 20.3 Study participation is voluntary. The information will be given in written form (ICF) as well as verbally by the investigator.
- **20.4** The subject's LAR will sign and date the ICF. The ICF will then be dated and signed by the investigator.
- **20.5** The investigator will retain the original of the documents. The subject's LAR will receive a copy of the ICF and if applicable, insurance terms and conditions.

#### 21.0 Adverse events and adverse device effects


The procedures to be performed under this protocol are considered to be of low risk since the glucose testing procedures will use residual samples which are remnants of neonatal blood collected as part of routine prescribed practice.

Due to the nature of this study, no adverse events (AE) are expected as per the following:

- 21.1 This study only includes residual ('left-over') samples of blood collected by standard, approved technique for prescribed tests.
- 21.2 No neonate will be exposed to any of the BGMS at any point; all study activities will be conducted in the institution's lab.
- **21.3** The samples will be de-identified in order to protect the confidentiality of the subjects. Confidentiality issues are mitigated due to the fact that the nursing staff overseeing the babies will not be informed of any study results, and samples will be de-identified prior to being given to the laboratory staff who perform study testing
- **21.4** Regardless of the above, any experience that the investigator considers to be an AE will be documented and reported immediately to Ascensia.

#### **21.5** Definition of Adverse Events

21.5.1 Adverse Event (AE): Adverse event refers to any untoward medical occurrence, inappropriate patient management decision, unintended disease or injury, or untoward clinical signs in subjects, users, or other persons, with any connection to to study related activities, whether or not related to the IVD medical device under investigation.

Protocol /CIP: GCA-PRO-2021-003-01 - Amendment 1

Ascensia Diabetes Care

Version: 14Oct2022


21.5.2 <u>Adverse Device Effect</u> (ADE or Adverse Effect): Any AE resulting from insufficient or inadequate instructions for use, installation, operation, or any malfunction of the IVD medical Device under investigation. This includes any AE resulting from use error or from unintentional misuse of the device.

- 21.5.3 Serious Adverse Event (SAE): Refers to an AE that led to any of the following:
  - a) death,
  - b) serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
    - 1) a life-threatening illness or injury, or
    - 2) a permanent impairment of a body structure or a body function including chronic diseases, or
    - 3) in-patient or prolonged hospitalisation, or
    - 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
  - c) fetal distress, fetal death, or a congenital abnormality or birth defect, including physical or mental impairment.
- 21.5.4 <u>Serious Adverse Device Effect</u> (SADE): Adverse device effect that has resulted in any of the consequences of an SAE.

#### 21.6 Adverse Event Classification

**Table 3. Classification of Adverse Events** (ISO 20916: 2019)

| Adverse Events | Non -device related | Device related | |
|---|---|---|---|
| | Applies to : Interventional Studies Sampling procedure causes direct harm to the subject | <ul> <li>Applies to:</li> <li>Interventional Studies: inaccurate test result leads to indirect harm to the subject.</li> <li>Sampling procedure causes direct harm to the subject</li> </ul> | |
| Non-Serious | Adverse event (includes all categories) | Adverse device effect | |
| Serious | Serious Adverse event (includes all categories that are serious) | Serious adverse device effect | |
| | | Anticipated | Unanticipated |
| | | Anticipated Serious adverse device effect | Unanticipated Serious adverse device effect |

#### 21.7 Adverse Event Reporting

- 21.7.1 AEs will be documented during this study by completing the AE Form. The Investigator or designee will sign and date an AE Form for each AE that is observed.
- 21.7.2 AEs will be evaluated by a member of the study staff and the PI. The nature of each event and date of onset, outcome, course, maximum intensity and action taken for treatment should be established. Details of any corrective treatment should be recorded on the AE Form.
- 21.7.3 Investigators should follow up on the status of any AE until the event has been resolved, or until the condition has stabilized.
- 21.7.4 The Investigator or designee will notify the Study Manager or Study Monitor within 24 hours of any SAE that occurred during the study. Ascensia will promptly review all information relevant to the safety of the investigational device.
- 21.7.5 Upon the receipt of a report of an SAE by the Ascensia Study Manager or Monitor, the report will be immediately forwarded to:



# 22.0 Handling and Reporting of Device Deficiencies

- **22.1** Any functional problems with the investigational BGMS will be considered a device deficiency and will be documented by the study staff and reported timely to Ascensia.
- **22.2** The study staff should be specific about describing the problem and the sequence of events that led to it. All information will be documented on the Data Deficiency Form, including the meter type, serial number, and test strip lot.
- **22.3** Malfunctioning BGMs will be replaced and this will be documented for device tracking.
- **22.4** All device deficiencies related to the identity, quality, durability, reliability, safety or performance of an investigational medical device shall be documented throughout the clinical investigation and appropriately managed by the sponsor.
- **22.5** Device deficiencies that did not lead to an AE but could have led to a medical occurrence shall be reported to the sponsor without delay.
- **22.6** All device deficiencies are to be reviewed and documented in writing whether they could have led to a SADE.

# 23.0 Vulnerable population

**23.1** While the samples will be taken from neonates, who are in the vulnerable population category, the procedure does not involve additional risk since the samples are residual with no additional sampling required.

**23.2** If the IRB determines consent is required, then proxy consent by an LAR shall be provided to protect the rights of the subject.

# 24.0 Suspension/Premature termination and Subject Withdrawal Criteria

- **24.1** In the event the study is prematurely suspended or terminated, the sponsor shall be notified as well as the IRB.
- **24.2** The subject's sample may be withdrawn from the study at the discretion of the Investigator.

# 25.0 Results Handling

Results of the study will not be shared with subjects. There is no plan for treating or following up with subjects based on the investigational results from this study.

# 26.0 Publication policy

- **26.1** The results will be published in regulatory databases, Clinicaltrials.gov and EUDAMED.
- 26.2 In general, for publication of data, the principles of GCP and Good Scientific Practice are respected. All manuscripts, abstracts or other modes of presentation arising from the results of the study must be reviewed and approved in writing by the sponsor in advance of submission. The sponsor's intention is neither to influence nor to prevent the publication of the study results to the medical and scientific community. The review is exclusively aimed at protecting the sponsor's proprietary information existing either at the date of commencement of the study or generated during the study. Details of the publication policy and related sponsor and principal investigator responsibilities are included in the clinical investigation agreement.


#### 27.0 Administration

All investigator and site staff communications regarding the study should be directed to the Ascensia Study Manager. If at any time questions or problems arise concerning the evaluation, please contact the Ascensia Study Manager at the telephone number listed below.



# 28.0 Bibliography

- 1. Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. *Pediatrics* 2011; 127: 575–79.
- 2. British Association of Perinatal Medicine. Identification and management of neonatal hypocycaemia in the full term infant. A BAPM framework for practice. 2017. https://www.bapm.org/resources/40-identification-and-management-of-neonatalhypoglycaemia-in-the-full-term-infant-2017 (accessed Sept 23, 2020).
- 3. CLSI. Point-of-Care Blood Glucose Testing in Acute and Chronic Care Facilities; Approved Guideline Third Edition. CLSI document POCT 12–A3. Wayne, PA: Clinical and Laboratory Standards Institute: 2013.
- 4. Draper, N.R. and Smith, H. (1998). *Applied Regression Analysis*, 3<sup>rd</sup> Ed., John Wiley and Sons, NY.
- 5. Harris DL, Weston PJ, Harding JE. Incidence of neonatal hypoglycemia in babies identified as at risk. *J Pediatr*. 2012;161:787-791.
- 6. ISO 15197: 2013. In vitro diagnostic test systems-requirements for blood glucose monitoring systems for self-testing in managing diabetes mellitus. Reference number ISO: 2013(E), Geneva: International Organization for Standardization; 2013.
- 7. ISO 20916: 2019. In vitro diagnostic medical devices—clinical performance studies using specimens fro human subjects—Good Study Practice. Geneva: International Organization for Standardization (ISO); 2019.
- 8. ISO 22870: 2016. Point-of-care testing (POCT)—requirements for quality and competence. Geneva: International Organization for Standardization (ISO); 2016.
- 9. Lucas A, Morley R, Cole TJ. Adverse neurodevelopmental outcome of moderate neonatal hypoglycaemia. *BMJ* 1988;297:1304–8.
- 10. Movalia MK, Ogino MT. Point of care glucose testing in neonatal hypoglycemia. *Point Care*. 2006;5:95–9.
- 11. Nuntnarumit P, Chittamma A, Pongmee P, Tangnoo A, Goonthon S. Clinical performance of the new glucometer in the nursery and neonatal intensive care unit. *Pediatr Int.* 2011;53:218–23.
- 12. Roth-Kleiner M, Stadelmann Diaw C, Urfer J, Ruffieux C, Werner D. Evaluation of different POCT devices for glucose measurement in a clinical neonatal setting. *Eur J Pediatr*. 2010;169:1387–95.
- 13. Rozance PJ, Hay WW. Hypoglycemia in newborn infants: features associated with adverse outcomes. *Biol Neonate*. 2006;90:74-86.


# **Appendix A - Instructions for Cleaning and Disinfecting Meters**

Study staff will clean and disinfect meters according to the UG instructions for HCPs.

#### **Health Care Professionals**

Health care professionals or persons using this system on multiple patients should follow the infection control procedure and the recommendations for prevention of blood-borne transmissible diseases approved by their facility.

The following disinfection solutions are recommended: 70% isopropyl alcohol, 6.0% sodium hypochlorite (full bleach), 0.6% sodium hypochlorite (diluted bleach), didecyldimethylammonium chloride (DDAC).

<u>NOTE:</u> Using cleaning and disinfecting solutions other than those recommended by the manufacturer could result in damage to system components. The cleaning and disinfecting directions provided should not cause any damage or degradation to the external case, buttons, or display.

<u>CAUTION</u>: Do not allow any solution to run into the meter through open areas, such as around the buttons or the meters test strip or data ports, such as USB port.

Blood glucose meters must be cleaned and disinfected by study staff before returning to Ascensia.

#### References

Protection of laboratory workers from occupationally acquired infections; approved guideline – third edition. CLSI document M29-A3. ISBN1-56238-567-4.

Rutala W, Weber D. Healthcare Infection Control Practices Advisory Committee. Guideline for disinfection and sterilization in healthcare facilities, 2008. Centers for Disease Control and Prevention.

# Appendix B - Instructions for Processing of Blood for the glucose analyzer

#### Processing of Neonatal Blood for laboratory glucose analysis

Once collected, process the microtainer tube for laboratory glucose analysis as follows:

- Label all tubes with the subject number using a Sharpie<sup>®</sup>-like marker.
- Gently invert the microtainer tube several times to mix the anticoagulant.
- Centrifuge the whole blood immediately to separate the plasma from the red blood cells. The centrifugation start time must occur within 10 minutes of the first meter blood test. The timing of all meter testing/centrifugation will be recorded on the appropriate CRF.
- It is recommended that after centrifugation, the plasma is transferred from the microtainer tube to a small clean tube or container with a cap. Ensure the tube is labeled and the cap is secured, and proceed with the site's laboratory glucose analyzer procedures.
- The plasma will be tested in duplicate with the laboratory analyzer within 60 minutes of the meter test. If greater than 60 minutes of the meter test, plasma samples may be refrigerated.
- Insufficient (or suspected to be insufficient) samples, missing samples, and other sample issues should be recorded in the CRF and on the glucose analyzer printout, as appropriate. If a sample is hemolyzed, record it in the CRF.

# **Appendix** C - Instructions for Tracking Accuracy and Precision of the Laboratory Glucose Analyzer

Procedure for Tracking Accuracy and Precision of Site Laboratory Analyzer

Performance of the Cobas 6000 will be assessed to ensure accuracy. Analyzer performance will be tracked by two methods: the Laboratory Analyzer QC procedure regularly applied by the clinical site, and the testing of serum controls provided by Ascensia.

The following are the procedures required for each method:

#### I. Laboratory Analyzer QC Procedure

The Cobas 6000 will be maintained and operated according to the instructions in the manufacturer's operating manual by the site's lab specifications/SOP previously reviewed by ADC. Before the study begins, the analyzer will be set up and the appropriate maintenance will be performed.

The site will perform glucose analyzer control tests in accordance with the site's quality control check procedures and requirements. Site staff will keep a log for the analyzer, including daily operational checks and maintenance.

#### II. Ascensia Serum Controls<sup>1</sup>

A set of three serum control levels will be provided to the investigator to document the performance of the Cobas 6000 at each BG level. These serum controls have been assayed by a method traceable to one proposed for use as a national glucose reference method.

#### Serum Control Testing Schedule:

- Pre-study: The controls will be assayed (singlet readings) on the Laboratory Analyzer for at least three runs prior to the assay of subject samples. The runs will occur over at least three days, if possible. The data will be sent to the Ascensia Study Manager, or designee, for review before the study begins.
- Once the study begins, serum control testing should be completed on each Analyzer on the Monday and Friday of the first week, and then on one day for each week that the study continues.
- Record all data on the CRF. One reading will be recorded for each control level (for a total of 3 readings per run).

<sup>&</sup>lt;sup>1</sup> Caution: The serum glucose traceability controls are human serum-based and must be handled using universal precautions.

#### Proper Handling of Ascensia Serum Controls

Ascensia completed the characterization of serum controls purchased from Bio-Techne® (formerly Bionostics). During the characterization, staff observed that sample stratification during thawing can occur if the control vials are not handled judiciously. The recommended procedure is as follows.

- Store the frozen controls in a -20C freezer upon arrival.
- Thaw the frozen control amber glass vials at 2-8°C for 2-3 days in the refrigerator. Each vial holds approximately 2.0 mL.
- Before opening, mix the vials well by gently inverting them at least 10 times.
- Prepare an aliquot of each level in capped microcentrifuge tubes. Cap tightly. We prefer Fisherbrand<sup>™</sup> Microcentrifuge 0.5mL tubes (PN 02-681-333) with O-ring seal caps (PN 02-681-358).
- Store any remaining control in the amber glass vials at 2-8°C.
- Before running a control sample on the laboratory analyzer, mix the aliquot tubes by gently inverting them.
- At the beginning of each day, remix the amber glass vials and refill the aliquot tubes. When not in use, store the aliquots at 2-8°C.
- The thawed control use life is two weeks. Discard all thawed control—aliquot tubes and amber glass vials—after two weeks.
- Since slow thawing for 2-3 days is recommended, it is advisable to keep an extra thawed set available for testing.

# **Appendix D - Instructions for Hematocrit Sample Preparation and Testing**

Staff will follow the instructions in the hematocrit reader user manual.

- 1. At least one microhematocrit tube, but preferably two, will be filled with residual capillary blood from each subject sample. One tube will be measured, and the result recorded on the form. The second tube is a backup and will be measured only if the first tube was not adequate for measurement, or is broken.
  - Ensure the tube setting on the HemataStat II<sup>TM</sup> is set to 0.5 mm ID (inner diameter).
  - Samples collected from residual capillary blood (heel-stick) will be collected in treated micro-hematocrit tubes.
- 2. Place a microhematocrit tube against the surface of the blood drop.
- 3. Fill the microhematocrit tube about halfway. Do not over-fill. Then immediately place one of the microhematocrit tube openings in the clay sealant. Press into the clay 2-3 times to make sure enough sealant is transferred.
- 4. Place the sealed microhematocrit tube into the Hematastat II<sup>TM</sup> micro-centrifuge. Note: it is very important to place the microhematocrit tube in centrifuge rotor with clay side down. Balance the rotor with another hematocrit tube containing water.
- 5. Click run to spin for the preset 60 seconds.
- 6. Measure hematocrit using the Hematastat reader or other hematocrit reader approved by the sponsor.
- 7. Summary of Instructions for the Hematastat reader:
  - After collection and centrifugation of hematocrit, place tube in the reader slot, with clay side to the left. Press enter to read.
  - Slide the marker on the reader to the exact line where the clay and red blood cells meet. Press enter to "enter interface: sealant/RBCs."
  - Then move the marker to the exact line where the red blood cells meet the plasma. Press enter to "enter interface: RBCs/plasma."
  - Slide the marker to the exact line where the plasma ends. Press enter to "enter interface: plasma/air."
  - The result in the display is the hematocrit percentage for that sample.
- 8. Record hematocrit result on the appropriate form.

# **Attachment 1 - CONTOUR NEXT User Guide**





# **Attachment 2 - CONTOUR PLUS ELITE User Guide**



